CLINICAL TRIAL: NCT03722108
Title: A Randomised Phase 2 Trial Assessing REGorafenib Combined With IRInotecan as Second-line Treatment in Patients With Metastatic Gastro-oesophageal Adenocarcinomas
Brief Title: Regorafenib Combined With Irinotecan as Second-line in Patients With Metastatic Gastro-oesophageal Adenocarcinomas
Acronym: REGIRI
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unfavorable benefit-risk balance in the experimental arm following the IDMC for intermediate efficacy and safety analysis
Sponsor: UNICANCER (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0110/1807; 2018-002374-46 (EudraCT Number)
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Adenocarcinoma of the Stomach; Adenocarcinoma of the Gastroesophageal Junction
Keywords: adenocarcinoma; gastro-oesophageal; regorafenib
MeSH Terms: conditions — Adenocarcinoma | interventions — regorafenib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regorafenib and Irinotecan (Experimental): Irinotecan 180 mg/m² on Day1 and Day 15 of a 4 week cycle combined with regorafenib 160 mg daily on Day2-8 and D16-22 of a 4 week cycle administered until progression of disease or unacceptable toxicity.
  Interventions: Combination Product: Regorafenib and Irinotecan
- Irinotecan (Active Comparator): Irinotecan 180 mg/m² on Day1 and Day 15 of a 4 week cycle administered until progression of disease or unacceptable toxicity
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Combination Product: Regorafenib and Irinotecan — Irinotecan (180 mg/m² on D1 and D15 of a 4-week cycle) combined with regorafenib (160 mg daily on D2-8 and D16-22 of a 4-week cycle) administered until progression of disease or unacceptable toxicity
  Other Names: STIVARGA; CAMPTO
  Arms: Regorafenib and Irinotecan
Drug: Irinotecan — Irinotecan (180 mg/m² on D1 and D15 of a 4-week cycle) administered until progression of disease or unacceptable toxicity
  Other Names: CAMPTO
  Arms: Irinotecan

SUMMARY:
Trial evaluating the efficacy of regorafenib combined with irinotecan compared to irinotecan alone in second-line treatment of patients with metastatic gastro-oesophageal adenocarcinomas.

DETAILED DESCRIPTION:
Comparative interventional prospective phase 2, randomised, open-label, multicentric trial comparing the combination of regorafenib and irinotecan (REGIRI) to irinotecan alone (IRI) as second line treatment of patients with metastatic gastro-oesophageal adenocarcinomas.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed a written informed consent form prior to any study specific procedures
2. Patients aged ≥18 years old
3. Histologically confirmed diagnosis of gastro-oesophageal adenocarcinomas: gastroesophageal junction (Siewert II and III) and gastric adenocarcinomas
4. Asymptomatic primary tumour
5. Metastatic disease
6. At least one target lesion (according to RECIST v1.1):

   * Unidimensionally measurable on cross-sectional imaging
   * In an area not previously irradiated
7. Disease progression after a fluoropyrimidine and platinum agent-based chemotherapy (5-fluorouracil or 5-fluorouracil prodrugs combined with cisplatin or oxaliplatin). For example, docetaxel combined with FOLFOX, PD-L1/PD-1 inhibitors combined with FOLFOX, LV5-FU2-cisplatin or 5-fluorouracil-cisplatin are acceptable prior therapies.
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
9. Life expectancy >3 months
10. Amylase ≤1.5 x upper limit of normal (ULN) and lipase ≤1.5 x ULN
11. Adequate liver function:

    * Total bilirubin ≤1.5 x ULN
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 x ULN (≤5 x ULN for patients with liver metastasis)
    * Alkaline phosphatase (ALP) ≤2.5 x ULN (≤5.0 x ULN for patients with liver or bone metastases)
12. Platelet count ≥100,000/mm³; haemoglobin (Hb) ≥9 g/dL; absolute neutrophil count (ANC) ≥1,500/mm³. The use of blood transfusion(s) to meet the inclusion criteria will not be allowed
13. International normalised ratio (INR) ≤1.5 x ULN and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤1.5 x ULN unless receiving treatment with therapeutic anticoagulation. Patients being treated with anticoagulant, e.g., heparin, are eligible if there is no evidence of an underlying abnormality with these parameters and if a close monitoring of at least weekly evaluations was performed until INR and PTT are stable based on a pre-dose measurement as defined by the local standard of care
14. Creatinine clearance (CLcr) ≥50 mL/min estimated by Cockcroft-Gault equation
15. Women of childbearing potential and men must agree to use adequate contraception during the study and for at least 3 months after the last study drug administration
16. Patients affiliated to the social security system

Exclusion Criteria:

1. Symptomatic brain metastases or carcinomatous meningitis
2. Bone-only metastasis
3. Known and documented UGT1A1 deficiency
4. History of Gilbert's syndrome
5. Previous or concurrent cancer with a distinct primary site, other than gastro-oesophageal cancer, within 5 years prior to randomisation (except for curatively treated cervical cancer in situ, non-melanoma skin cancer, and superficial bladder tumours)
6. Persistent proteinuria >3.5 g/24 h measured by urine protein-creatinine ratio from a random urine sample (grade ≥3, NCI-CTCAE v 5.0)
7. Interstitial lung disease with ongoing signs and symptoms at inclusion
8. Known hypersensitivity to any of the study drugs, study drug classes, or excipients
9. Non-healing wound, non-healing ulcer, or non-healing bone fracture
10. Patients with evidence or history of any bleeding diathesis, irrespective of severity
11. Any haemorrhage or bleeding event grade ≥3 (NCI-CTCAE v.5.0) within 4 weeks before starting of the study treatment
12. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 month before starting the study treatment (except for adequately treated catheter-related venous thrombosis occurring more than one month before the start of study medication)
13. Previous major surgical procedure, significant traumatic injury, or radiotherapy within the 4 weeks before inclusion
14. Uncontrolled hypertension (systolic blood pressure >140 mmHg or diastolic pressure >90 mmHg) despite optimal medical management. Congestive heart failure: New York Heart Association (NYHA) ≥ class 2
15. Unstable angina (angina symptoms at rest), new-onset angina (that started within the last 3 months)
16. Myocardial infarction less than 6 months before starting the study treatment
17. Uncontrolled cardiac arrhythmias
18. History of epileptic seizures requiring long-term anticonvulsant therapy
19. History of organ transplantation with use of immunosuppression therapy
20. Ongoing bacterial or fungal infection (grade >2 by NCI-CTCAE v.5.0)
21. Known history of human immunodeficiency virus (HIV) infection
22. Active hepatitis B or C, or chronic hepatitis B or C requiring treatment with antiviral therapy
23. Use of CYP3A4 inducers or inhibitors
24. Pregnant or breast-feeding women
25. Bowel malabsorption or extended bowel resection that could affect the absorption of regorafenib, occlusive syndrome, inability to take oral medications
26. Inflammatory bowel disease with chronic diarrhoea
27. Participation in another clinical trial within the 30 days before inclusion
28. Concurrent treatment with another investigational product or anticancer therapy (other than irinotecan or regorafenib)
29. Concomitant treatment with hypericum or live attenuated vaccines
30. Gastro-intestinal fistula or perforation
31. Person kept in detention or incapable of giving consent
32. Patient unwilling or unable to comply with the medical follow-up required by the study because of geographic, social, or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of regorafenib combined with irinotecan versus irinotecan alone in terms of overall survival (OS) | expected duration of 10 months from randomisation
  Time duration from randomisation to time of death of any cause. If a patient is alive at the database cut-off date, then the patient will be censored at the last date of follow-up.

SECONDARY OUTCOMES:
To compare the efficacy of regorafenib combined with irinotecan versus irinotecan alone in terms of the overall survival rate | 6 and 12 months from randomisation
  Overall survival rates at 6 and 12 months
To compare the efficacy of regorafenib combined with irinotecan versus irinotecan alone in terms of the progression-free survival (PFS) | expected duration of 6 months from randomisation
  Time duration from randomisation to time of first event (locoregional or distant relapse or progression, second malignancy, death from any cause).
To evaluate the efficacy of regorafenib combined with irinotecan versus irinotecan alone in terms of the progression-free survival rate | 6 and 12 months from randomisation
  Progression-free survival rates at 6 and 12 months
To evaluate the efficacy of regorafenib combined with irinotecan versus irinotecan alone in terms of the disease control rate (DCR) | expected duration of 6 months from randomisation
  Percentage of patients with complete response, partial response or stable disease as best response at the database cut-off date
To evaluate the efficacy of regorafenib combined with irinotecan versus irinotecan alone in terms of the objective response rate (ORR) | expected duration of 6 months from randomisation
  Percentage of patients with complete response or partial response
To compare treatment-related toxicity | expected 30 days after last study treatment administration
  Frequency and severity of adverse events assessed by NCI-CTCAE v5.0
To compare the effect of treatment on quality of life | expected 30 days after last study treatment administration
  Evaluation of quality of life with EORTC quality of life questionnaire for cancer patients (QLQ-C30)
To compare the effect of treatment on quality of life related to gastro-oesophageal cancer | expected 30 days after last study treatment administration
  Evaluation of quality of life with EORTC quality of life specific questionnaire for gastro-oesophageal tumours (QLQ-OG25)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle SAMALIN-SCALZI, MD, Principal Investigator — Institut du Cancer Montpellier
Locations (27):
- France (27):
  - Institut de Cancérologie de l'Ouest-Paul Papin, Angers
  - Hôpital Morvan, Brest
  - Clinique de Flandre, Coudekerque-Branche
  - Centre Georges François Leclerc, Dijon
  - Hôpital Franco-Britannique, Levallois-Perret
  - Hopital Claude Huriez - CHU Lille, Lille
  - CHU Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Hopital de la Timone, Marseille
  - Institut Paoli Calmette, Marseille
  - Institut du Cancer Montpellier, Montpellier
  - Centre de Cancérologie du Grand Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hopital Europeen Georges Pompidou, Paris
  - GH Diaconesses Croix Saint-Simon, Paris
  - CH Saint Jean, Perpignan
  - CHU de Poitiers, Poitiers
  - CH Annecy Genevois, Pringy
  - Institut Jean Godinot, Reims
  - Hopital Robert Debre, Reims
  - Hopital Charles Nicolle, Rouen
  - CHP Saint Grégoire, Saint-Grégoire
  - Institut de Cancérologie de l'Ouest-René Gauducheau, Saint-Herblain
  - CH Saint Malo, St-Malo
  - Centre Paul Strass, Strasbourg
  - CHRU Tours, Tours
  - CHU Nancy - Hôpital Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level, they will be part of the study database including all enrolled patients